CLINICAL TRIAL: NCT05462457
Title: Prospective, Multicentric Registry Study Evaluating the False-negative Rate of Targeted Axillary Dissection (TAD) in Primary Breast Cancer With Initially ≥ 3 Suspicious Lymph Nodes Under Neoadjuvant Systemic Therapy (SenTa 2)
Brief Title: TAD in Primary Breast Cancer With Initially ≥ 3 Suspicious Lymph Nodes
Acronym: SenTa2
Status: Recruiting | Type: Observational
Sponsor: Kliniken Essen-Mitte (Other)
Responsible Party: Sponsor
Other Study IDs: Version 1.0_16.08.2021
Record Dates: First submitted 2022-07-14; First posted 2022-07-18 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer; Node-positive Breast Cancer
Keywords: Targeted axillary dissection; TAD; False-negative rate
MeSH Terms: conditions — Breast Neoplasms | interventions — DAT protocol 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Paraffin-embedded lymph nodes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Targeted axilllary dissection (TAD) followed by axillary lymph node dissection (ALND) — Intraoperative excision of TAD lymph nodes followed by ALND in the same surgical session or secondary surgical intervention

SUMMARY:
Due to high pathological complete remission (pCR) rates in both breast and lymph nodes (ypT0/Tis, ypN0) following neoadjuvant systemic therapy (NST) in many patients with initially clinically node-positive (cN+) breast cancer, the standard treatment of the axilla has changed from axillary lymph node dissection (ALND), which is associated with high morbidity, to less invasive, surgical approaches. In several studies, targeted axillary dissection (TAD) has presented with false-negative rates (FNRs) less than 5%, however, in patients with high initial lymph node involvement (≥ 3 clinically suspicious lymph nodes) TAD has not been thoroughly investigated.

The present prospective registry study aims to evaluate the FNR of TAD in patients with ≥ 3 initially suspicious lymph nodes and clinically node-negative status (ycN0) after NST in comparison to ALND.

DETAILED DESCRIPTION:
Patients with triple-negative breast cancer (TNBC) or human epidermal growth factor receptor 2 (HER2) positive breast cancer achieved pCR rates of 50-70% following NST. In the multicenter prospective SenTa study (NCT03102307), the axillary pCR rate after the end of NST in 473 initially cN+ patients was 60.3%. Therefore, less invasive surgical techniques have been investigated to avoid the morbidity associated with ALND. One of these minimally invasive methods called TAD involves the combined intraoperative excision of the pre-NST marked most suspicious lymph node (target lymph node, TLN) and sentinel lymph nodes (SLNs). In a pooled analysis of 13 studies including 521 patients who had undergone TAD, the FNR of TAD was 5.2%.

The FNR of TAD in breast cancer patients with high initial lymph node (LN) involvement (≥ 3 clinically suspicious LNs) has so far hardly been investigated. In a very small cohort, a FNR of 0% was obtained for patients with 1-3 suspicious LNs (cN1, n = 10), 33% for patients with 4-9 suspicious LNs (cN2, n = 3) and 100% for patients with 10 or more suspicious LNs (cN3, n = 2). In addition, patients with high lymph node involvement are often excluded from some larger studies evaluating TAD or other axillary surgical approaches. In consequence, the FNR of TAD LNs in comparison to LNs obtained during ALND in the patient group with ≥ 3 clinically positive LNs needs to be evaluated in a larger cohort, since extensive initial LN involvement is associated with a higher probability that a false-negative result of TAD could cause one or more involved LNs to be left in the axilla, if only TAD and not ALND is performed.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent form
* female/male patient aged ≥ 18 years
* clinical (c) tumor stage T1-4c, bilateral breast cancer and multifocal tumor allowed
* invasive breast cancer confirmed by core biopsy
* clinically node positive (cN+) (by means of axillary ultrasound or other imaging methods) with ≥ 3 clinically suspicious lymph nodes
* biopsy-proven axillary lymph node involvement
* marking (e.g. with a clip, magnetic seed, carbon suspension) of the clinically suspicious lymph node(s) before the start of NST
* without distant metastases
* indication for NST including chemotherapy
* TAD + ALND planned
* at least 7 lymph nodes (TAD + ALND) planned for histological analysis

Exclusion Criteria:

* cN0 or cN+ with ≤ 2 clinically suspicious lymph nodes
* patients without indication for NST or NST < 12 weeks
* NST without chemotherapy
* adjuvant/ neoadjuvant therapy already started prior to inclusion in the study
* patients for whom only ALND is planned
* ycN+ (by means of axillary ultrasound or other imaging methods)
* recurrent breast cancer
* larger surgery of the breast (starting from quadrant resection) or the axilla prior to the study
* previous radiotherapy of the breast or axilla
* inflammatory breast cancer
* extramammary breast cancer
* pregnant women
* not able to undergo surgery
* inability to understand the purpose of the clinical study or to comply with study conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary breast cancer and ≥ 3 (initially) clinically positive lymph nodes with an indication for NST and in whom TAD + ALND is planned when ycN0 status is achieved after the end of NST.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-03-07 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2032-03 (Estimated)

PRIMARY OUTCOMES:
False-negative rate (FNR) of TAD in patients with ycN0 status | Postoperatively immediately after histopathological evaluation of LNs
  The FNR of TAD is calculated as the number of patients with histologically negative TAD lymph nodes (LNs) who were found to have positive LNs in the ALND specimen, divided by the total number of patients with positive LNs.

SECONDARY OUTCOMES:
Detection rate of preoperative ultrasound | Preoperatively
  Preoperative detection rate (DR) of initially marked target lymph nodes (TLNs) on ultrasound images after the end of NST
Localization of TLNs | Preoperatively or during NST
  Successful localization with e.g. wire, magnetic marker, or reflector clip of the marked TLNs
Detection rate of TAD | At the time of surgery
  Successful intraoperative identification of at least one SLN and one TLN, including cases with TLN = SLN
Detection rate of target lymph node biopsy (TLNB) | At the time of surgery
  Successful intraoperative identification of TLN(s)
Detection rate of sentinel lymph node biopsy (SLNB) | At the time of surgery
  Successful intraoperative identification of SLN(s)
FNR of TLNB | Postoperatively immediately after histopathological evaluation of LNs
  The FNR of TLNB is calculated as the number of patients with histologically negative TLNs who were found to have positive SLNs and/or positive LNs in the ALND specimen, divided by the total number of patients with positive LNs.
FNR of SLNB | Postoperatively immediately after histopathological evaluation of LNs
  The FNR of SLNB is calculated as the number of patients with negative SLNs who were found to have positive TLNs and/or positive LNs in the ALND specimen, divided by the total number of patients with positive LNs.
FNR of preoperative ultrasound | Postoperatively immediately after histopathological evaluation of LNs
  False-negative is defined as preoperative ycN0 status on axillary ultrasound images and pathological ypN+ after surgery
Rate of local recurrence | 5 years after surgery, interim analysis: 2 years after surgery
  Proportion of patients with ipsilateral or contralateral recurrence in the breast and/or axilla occurring at any time after surgery.
Rate of distant recurrence | 5 years after surgery, interim analysis: 2 years after surgery
  Proportion of patients with distant recurrence occurring at any time after surgery.
Invasive disease-free-survival (iDFS) | 5 years after surgery, interim analysis: 2 years after surgery
  iDFS is calculated as the time from surgery to the occurrence of either local recurrence, distant recurrence, second malignant disease (breast or different origin), or death from any cause.
Overall survival (OS) | 5 years after surgery, interim analysis: 2 years after surgery
  OS is calculated as the time from surgery to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Sherko Kuemmel, Prof. Dr., Study Chair — Breast Unit, Kliniken Essen-Mitte, Essen, Germany; Mattea Reinisch, Dr., Study Chair — Breast Unit, Kliniken Essen-Mitte, Essen, Germany
Locations (1):
- Kliniken Essen-Mitte (KEM), Essen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kuemmel S, Heil J, Rueland A, Seiberling C, Harrach H, Schindowski D, Lubitz J, Hellerhoff K, Ankel C, Grasshoff ST, Deuschle P, Hanf V, Belke K, Dall P, Dorn J, Kaltenecker G, Kuehn T, Beckmann U, Potenberg J, Blohmer JU, Kostara A, Breit E, Holtschmidt J, Traut E, Reinisch M. A Prospective, Multicenter Registry Study to Evaluate the Clinical Feasibility of Targeted Axillary Dissection (TAD) in Node-positive Breast Cancer Patients. Ann Surg. 2022 Nov 1;276(5):e553-e562. doi: 10.1097/SLA.0000000000004572. Epub 2020 Nov 4. PMID 33156057